CLINICAL TRIAL: NCT03711019
Title: Cognitive Outcomes and the Response/Remission Efficacy of Convulsive Therapies During Continuation: CORRECT-C Trial
Brief Title: Efficacy of Convulsive Therapies During Continuation
Acronym: CORRECT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of British Columbia (Other); Ontario Shores Centre for Mental Health Sciences (Other); Brain Canada (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head and Co-Director, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 022-2018
Record Dates: First submitted 2018-10-12; First posted 2018-10-18 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Depression; Bipolar Depression; Unipolar Depression; Treatment Resistant Depression
Keywords: Magnetic Seizure Therapy; Electroconvulsive Therapy
MeSH Terms: conditions — Depression; Bipolar Disorder; Depressive Disorder; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: The study will involve a parallel-group clinical trial with three treatment arms conducted at the Centre for Addiction and Mental Health (CAMH) in Toronto, ON, Ontario Shores Centre for Mental Health Sciences in Whitby, ON and UBC Hospital in Vancouver, BC.
  The investigators plan to enroll up to 105 participants to ensure 70 participants receive a complete course of continuation therapy following MST, RUL-UB ECT, or bitemporal ECT and anticipate enrolling up to 60 participants who will receive an acute course of bitemporal ECT as part of our secondary exploratory outcome over 48 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Individuals blinded to their acute course of treatment will continue to receive the convulsive therapy to which they responded in in a blinded fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Magnetic Seizure Therapy (MST) (Experimental): MST treatments will be administered using the MagPro MST with Cool TwinCoil.
  Interventions: Device: Magnetic Seizure Therapy (MST)
- RUL-UB ECT (Active Comparator): ECT treatments will be administered using the MECTA spECTrum 5000Q or MECTA Sigma
  Interventions: Device: RUL-UB ECT
- Bitemporal ECT (Active Comparator): ECT treatments will be administered using the MECTA spECTrum 5000Q or MECTA Sigma
  Interventions: Device: Bitemporal ECT

INTERVENTIONS:
Device: Magnetic Seizure Therapy (MST) — MST treatment will be administered using the MagPro MST with a Cool TwinCoil over the frontal cortex in the midline position using 100 Hz stimulation. Seizure threshold will have been determined during the first treatment session following a standard established protocol in the context of CREST-MST or CORRECT-BD. Treatment in the continuation phase will be administered at the same stimulus dose as the last treatment in acute phase.
  This will be performed under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes.
  Other Names: MST
  Arms: Magnetic Seizure Therapy (MST)
Device: RUL-UB ECT — In the RUL-UB ECT arm treatment, the MECTA spectrum 5000Q or MECTA Sigma machine will be used, which are FDA approved devices used for providing standard-of-care clinical ECT treatments. Seizure threshold will have been determined during the first treatment session following a standard established protocol in the context of CREST-MST or CORRECT-BD. Treatment in the continuation phase will be administered at the same stimulus dose as the last treatment in acute phase.
  This will be performed under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes.
  Arms: RUL-UB ECT
Device: Bitemporal ECT — Bitemporal ECT treatments will be administered using the MECTA spECTrum 5000Q or MECTA Sigma, which are FDA approved devices used for providing standard-of-care clinical ECT treatments. Bitemporal ECT will be administered at 1.5 times seizure threshold according to standard clinical practice. Treatment in the continuation phase will be administered at the same stimulus dose as the last treatment in acute phase.
  This will be performed under the effect of anesthesia. The treatment procedure is approximately 10 minutes, followed by a recovery period of approximately 30 minutes.
  Other Names: ECT
  Arms: Bitemporal ECT

SUMMARY:
This trial aims to assess the efficacy and tolerability of Magnetic Seizure Therapy (MST) and two different forms of electroconvulsive therapy (ECT) in sustaining response during and after a course of continuation treatment.

DETAILED DESCRIPTION:
The study will involve a parallel-group clinical trial with three treatment arms conducted at the Centre for Addiction and Mental Health (CAMH) in Toronto, ON, Ontario Shores Centre for Mental Health Sciences in Whitby, ON and University of British Columbia (UBC) Hospital in Vancouver, BC. It will include participants who are classified as responders or remitters in the CREST-MST (NCT03191058) trial, the CORRECT-BD (NCT03641300) trial and individuals responding to bitemporal ECT after participating in either of the above trials, who qualify for a continuation course of convulsive therapy to prevent relapse of depression. Individuals blinded to their acute course of treatment will continue to receive the convulsive therapy to which they responded in in a blinded fashion. Continuation treatments will be scheduled according to a modified version of the Symptom-Titrated Algorithm-based Longitudinal ECT (STABLE) algorithm. STABLE includes an initial four week period of ECT delivered on a fixed schedule (once or twice per week), and then transitions to a symptom-driven schedule whereby ECT is delivered between zero and two times per week based on the patient's weekly Hamilton Rating Scale for Depression (HRSD-24) outcomes during weeks five to 24.

Further, this trial will also include non-responders to MST or right unilateral ultrabrief pulse ECT (RUL-UB ECT) from CREST-MST or CORRECT-BD, who are switched to bitemporal ECT based on their clinical indication. They will receive bitemporal ECT on an acute basis, i.e. 2 - 3 times per week. If their symptoms respond or remit with bitemporal ECT, they will also be offered a continuation course of bitemporal ECT as part of this trial and will be followed in the same manner as those receiving MST or RUL-UB ECT.

ELIGIBILITY:
Participants in the Acute Phase (bitemporal ECT) will have already met the diagnostic criteria and severity eligibility criteria specified in the protocols of CREST-MST and CORRECT-BD.

At the time of recruitment, participants in the Continuation Phase (MST, RUL-UB ECT, Bitemporal ECT) will meet the following eligibility criteria:

Inclusion Criteria:

1. are inpatients or outpatients;
2. are voluntary and competent to consent to treatment and research procedures according to ECT/MST attending psychiatrist;
3. have met diagnostic criteria as assessed by MINI V6.0 in CREST-MST or CORRECT-BD
4. are 18 years of age or older
5. achieve remission defined as HRSD-24 < 10 and a > 60% decrease in scores from baseline on two consecutive ratings OR achieve response on HRSD-24 defined as a 50% reduction in symptoms from baseline;
6. are considered to be appropriate to receive convulsive therapy as assessed by an ECT attending psychiatrist and a consultant anaesthesiologist
7. are agreeable to keeping their current antidepressant treatment constant during the intervention;
8. are likely able to adhere to the intervention schedule;
9. meet the MST safety criteria;
10. If a woman of child-bearing potential: is willing to provide a negative pregnancy test and agrees not to become pregnant during trial participation.

Exclusion Criteria:

1. have a concomitant major unstable medical illness;
2. are pregnant or intend to get pregnant during the study;
3. have probable dementia based on study investigator assessment;
4. have any significant neurological disorder or condition likely to be associated with increased intracranial pressure or a space occupying brain lesion, e.g., cerebral aneurysm;
5. present with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, rheumatoid arthritis requiring high dose prednisone, or Cushing's disease);
6. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
7. require a benzodiazepine with dose greater than lorazepam 2 mg/day or equivalent or any anticonvulsant due to the potential of these medications to limit the efficacy of both MST and ECT;
8. are unable to communicate in English fluently enough to complete the neuropsychological tests;
9. have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Difference in HRSD-24 Scores between MST and RUL-UB at 6 months | 6 months
  Hamilton Rating Scale for Depression (24-item version):
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-76 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
  Non-inferiority trials such as this proposed study specify a non-inferiority margin, with a tolerance of 3.9 points denoting equivalence between the two treatments when the efficacy of MST can be concluded to be not more than 3.9 points on the HRSD-24 at the endpoint of treatment.
Cognitive adverse effects as indexed by the Autobiographical Memory Test (AMT) | 6 months
  Autobiographical Memory Test:
  * Interviewer-rated measure with 10 items that indexes autobiographical memory recall and specificity.
  * The binary outcome is defined as a worsening of > 25% on the AMT total score.

SECONDARY OUTCOMES:
Differences in relapse status between MST, RUL-UB ECT and bitemporal ECT | 6 months
  The secondary exploratory endpoint will investigate the differences between MST, RUL-UB ECT and bitemporal ECT on relapse status among participants during and after a course of continuation convulsive therapy.
Differences in HRSD-24 scores between MST, RUL-UB ECT and bitemporal ECT | 6 months
  Hamilton Rating Scale for Depression (24-item version):
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-76 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)
  A further endpoint will explore the difference on HRSD in those that receive MST, RUL-UB ECT and bitemporal ECT.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (3):
- Canada (3):
  - UBC Hospital, University of British Columbia (UBC), Vancouver, British Columbia
  - Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health, Toronto, Ontario
  - Ontario Shores Centre for Mental Health Sciences, Whitby, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research